CLINICAL TRIAL: NCT06359405
Title: Evaluation of Nursing Students' Crisis Management Skills in Medication Safety Simulation: A Randomized Controlled Study
Brief Title: Evaluation of Nursing Students' Crisis Management Skills in Medication Safety Simulation
Acronym: RCS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Seda Tugba Baykara Mat, Asst. Prof., University of Beykent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UBeykentUni
Record Dates: First submitted 2024-04-02; First posted 2024-04-11 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Nurse
Keywords: Nursing students; Medical Errors; Crisis management; Randomized Controlled Trial; Simulation Training

STUDY DESIGN:
Intervention Model Description: This study was planned as a randomized controlled study to evaluate the crisis management skills of student nurses in drug safety simulation.
Who Masked: Participant
Masking Description: The researchers declare that the data obtained from randomly formed groups will be numbered and entered into the statistical analysis program to hide the identity information and that two researchers will be assigned during the entry.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Working group (Experimental): The intervention will take place by presenting the simulation program to the working group.
  Interventions: Behavioral: drug safety simulation
- Control group (No Intervention): The control group will receive standard nursing education but not additional intervention.

INTERVENTIONS:
Behavioral: drug safety simulation — The intervention's purpose is to develop a simulation program to increase nursing students' crisis management skills regarding medication safety. This simulation program will provide students with the opportunity to develop skills in recognizing, evaluating, and effectively intervening in medication errors in real-world scenarios.
  The simulation program will include interactive case scenarios, virtual patients, and simulation sessions led by an instructor providing feedback to students. Also, medicine Learning materials covering preventing, recognizing, and correcting errors will also be provided.
  Arms: Working group

SUMMARY:
This study aims to objectively evaluate student nurses' crisis management skills in drug safety simulation and examine an effective intervention to improve these skills through a randomized controlled study. The research aims to provide important findings that will contribute to the determination of strategies to increase the competencies of student nurses in the fields of drug safety and crisis management.

Research Hypotheses:

H1: The application of drug safety simulation has an effect on the crisis management skill level of nursing students.

The aim of the intervention is to develop a simulation program to enhance nursing students' crisis management skills in drug safety. This simulation program will provide students with the opportunity to recognize, assess, and effectively intervene in medication errors in real-world scenarios.

The simulation program will include interactive case scenarios, virtual patients, and simulation sessions led by an instructor providing feedback to students. Additionally, learning materials covering topics such as prevention, recognition, and correction of medication errors will be provided

DETAILED DESCRIPTION:
The population and sample of the study have been calculated:

Number of 3rd and 4th-grade students: 70+71=141

Randomization: All 3rd-and 4th-grade students were included in the sample, and an independent statistician randomized them. Randomization will be done using the simple random sample selection table from the random.org website.

Control Group and Study Group: The research will use a randomized controlled trial design. Participants will be randomly assigned to two groups:

Control Group: The control group will receive standard nursing education and will not receive any additional intervention on drug safety and crisis management topics.

Study Group: The study group will participate in the simulation program and will receive the intervention designed to improve drug safety and crisis management skills.

The intervention will be implemented by providing the simulation program to the study group. The control group will receive standard nursing education but not additional intervention.

Data Collection for Post-test: Following the intervention phase, final test data will be collected from the participants.

Bias Prevention: Data from randomly generated groups will be anonymized with numbers during the research process, and entry into the statistical analysis program will be conducted in this way. Two researchers will be assigned during data entry.

Structured student introduction form: It consists of 6 questions regarding age, gender, economic status, and crisis-related experiences.

Crisis Management Scale: The scale aims to determine the approaches of school administrators to crisis management. The scale consists of 6 sub-dimensions and 45 items. The Cronbach's alpha coefficient of the Crisis Management Scale for nurse administrators is 0.85. In the study conducted with nurse administrators, after examining the internal consistency of the CMS, a reliability value of α = 0.754 was found.

Data Collection: The planned stages of data collection are listed below.

Implementation of the structured student introduction form Ensuring randomization Collection of initial test data Simulation application to the experimental group, conventional teaching method to the control group Collection of final test data

Intervention Content: The intervention aims to develop a simulation program to enhance nursing students' crisis management skills in drug safety. This simulation program will allow students to recognize, assess, and effectively intervene in medication errors in real-world scenarios. The program will include interactive case scenarios, virtual patients, and simulation sessions led by an instructor who provides student feedback. Additionally, learning materials covering topics such as prevention, recognition, and correction of medication errors will be provided.

Duration of the Intervention: The simulation program will be implemented in two stages for participants. The durations set for each stage are as follows:

Pre-test: Nursing students will take a pre-test on drug safety and crisis management topics before starting the simulation program. This test will be used to determine the students' baseline levels. The completion of the pre-test is estimated to take approximately 1 hour.

Simulation Program: The simulation program will be provided to students over several weeks. During this time, students are expected to participate in simulation sessions at specific time intervals and review educational materials on drug safety.

A detailed scenario will be used in this process. Expected behaviors in this scenario form; Knowledge, Skills and Behaviors Required Before the Scenario Knowledge - Explains the importance of drug safety.

* Knows the 8 truths in drug applications.
* Explains patient and employee safety in drug applications
* Explains the term Crisis Management
* Knows crisis management techniques Skill - Apply medication safety procedures
* Takes safety precautions in drug applications
* Applies the 8 truths in drug administration
* Manage the process during and after a crisis
* Uses crisis management techniques Behavior - Believes that medication safety is a key concept in patient and employee safety
* Believes in the necessity of safety precautions in drug administration
* Reflects the 8 truths in medication practices to care.
* Applies crisis management techniques
* Cold-blooded and cooperative behaviors will take place in the crisis management process.

Script Summary Your scenario takes place in the internal medicine ward of a hospital. A 69-year-old patient was admitted to the ward with complaints of dizziness, headache and general condition disorder. The patient was admitted from the emergency room. First intervention was made. The patient's anamnesis was tried to be taken quickly (this is how the nurse expresses it when delivering the patient). The patient has a spouse with him/her. Both the patient and his/her spouse are open to communication. You see the patient in the room for the first time. You are expected to initiate communication with the patient and perform the relevant nursing interventions.

It will include Patient Demographic Data, Standardized Patient / Simulator Features, Roles in the Simulation, and Pre-Information objectives.

Script Process Timing, Simulator Activities Expected Interventions Tips will be followed by focus group discussions using the debriefing session guide (PEARLS) to assess the alignment with the expected outputs in the Simulation Process Evaluation step.

Post-test: After completing the simulation program, students will take a post-test. This test will evaluate the student's progress in drug safety and crisis management skills following the simulation program.

The cris management scale will be used in pre and post tests.

Statistical Analysis of the Data: The data obtained in the research will be analyzed using the SPSS (Statistical Package for Social Sciences) for Windows 25.0

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Be registered in the nursing department
* Continuing formal education
* Having taken a Management course in Nursing

Exclusion Criteria:

* Being enrolled in a different program

  * Change of department/school
  * The student has a desire to leave the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-02 (Estimated)

PRIMARY OUTCOMES:
The effect of drug safety simulation application on the crisis management skill level of nursing students. | 3 Months
  The scale items are designed to make it easier for managers to answer:
  Before the crisis, During the crisis and Aftermath of the crisis The questionnaire was presented in three separate sections. In order to determine the crisis management approaches of nurse managers The answers given to the statements in the PBS used in the research are 5-point Likert type, The score ranged from 1 to 5 points from never to always. Accordingly;
  1. Never
  2. Very rare
  3. Occasionally
  4. Most of the time
  5. Always. 50 In addition, the mean scores of the sub-dimensions of the PBS; 1.00-1.79 points range is very negative 1.80-2.59 points is negative 2.60- 3.39 points in the range of 2.60- 3.39 points, medium level 3.40-4.19 points is positive A score between 4.20-5.00 is considered very positive

CONTACTS AND LOCATIONS:
Overall Officials: Seda Baykara Mat, Dr., Study Director — Asst. Prof.

IPD SHARING:
Plan to Share IPD: No
The information obtained from this study will be used entirely for research purposes and personal information will be kept confidential.